CLINICAL TRIAL: NCT03017014
Title: Assessing Long-term Safety and Effectiveness of Adalimumab for Treating Children and Adolescents With Crohn's Disease in Real Life Conditions-LEA
Brief Title: A Study to Assess Safety and Effectiveness of Adalimumab for Treating Children and Adolescents With Crohn's Disease in Real Life Conditions
Acronym: LEA
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-759
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Adalimumab; Humira®
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric participants receiving adalimumab: Pediatric participants receiving adalimumab for CD in real-life conditions.

SUMMARY:
The primary objective of this study is to evaluate long-term effectiveness of adalimumab in pediatric participants starting a treatment for Crohn's disease in real life conditions, namely to describe the time to loss of clinical benefit in a time to event approach. Main secondary objectives are to describe growth and pubertal development and to describe long-term safety. The participants will be followed-up up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* With confirmed diagnosis of Crohn's disease
* Adalimumab-naïve patient (a patient having received an anti-TNF other than adalimumab may enter the study)
* Starting a treatment with adalimumab
* Guardian capable of and willing to grant authorization for use/disclosure of data collected and patient able to comply with the requirements of the study protocol.

Exclusion Criteria:

* Participants with a history of treatment with adalimumab
* Participants enrolled in a concomitant interventional clinical trial.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants are children and adolescents with Crohn's disease
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Time to loss of clinical benefit | Up to 12 years
  Loss of clinical benefit will be defined as one of the following:
  * Loss of efficacy leading to adalimumab discontinuation or
  * Introduction / reinforcement of other immunosuppressants (ratio dose/weight) or
  * Introduction / reinforcement of corticosteroids (ratio dose/weight; reinforcement of corticosteroids are allowed within the 4 first months after start of adalimumab)
  * Introduction of enteral nutrition
  * CD-related surgery, discontinuation of adalimumab due to adverse event, death.

SECONDARY OUTCOMES:
Proportion of participants with dose escalation (dose and/or frequency of injections) | Up to 12 years
  Dosing and/or frequency of injections is monitored to assess dose escalation.
Median percent change from baseline in C-reactive protein (CRP) | From Month 0 to 12 years
  The median percent change from baseline in CRP is assessed at each time point.
Median percent change from baseline in calprotectin | From Month 0 to 12 years
  The median percent change from baseline in calprotectin us assessed at each time point.
Change from baseline in weighted Pediatric Crohn's Disease Activity Index (PCDAI) | From Month 0 to 12 years
  The Pediatric Activity Index (PCDAI) has become the standard outcome measure in pediatric Crohn's disease (CD) clinical research. The Weighted Pediatric Crohn's Disease Activity Index (wPCDAI) was developed to add weight to the items in the PCDAI and make it more feasible. In the wPCDAI, growth velocity, abdominal examination, and hematocrit are removed. The wPCDAI score can range from 0-125, with higher signifying severe disease activity.
Change in wPCDAI >= 37.5 | From Month 0 to 12 years
  A change in wPCDAI >= 37.5 indicates improvement.
Incidence rate of CD-related hospitalizations | Up to 12 years
  Hospitalization will be determined from the health care utilization information.
Rate of clinical remission | Up to 12 years
  Clinical remission is weighted PCDAI < 12.5 or Harvey-Bradshaw index (HBI) <5. Rate of clinical remission will be described at each time point
Proportion of participants achieving mucosal healing at each time point | Up to 12 years
  Mucosal healing is assessed using SES-CD score (0 or 1).
Proportion of participants with steroid-free clinical remission at each time point | Up to 12 years
  The proportion of participants with steroid-free clinical remission is assessed at each time point.
Change in weight z-score | From Month 0 to 12 years
  Growth is assessed by monitoring changes in weight z-score.
Median percent change from baseline in high sensitivity C-reactive protein (hs-CRP) | From Month 0 to 12 years
  The median percent change from baseline in hs-CRP is assessed at each time point.
Assessing Mucosal healing | Up to 12 years
  Mucosal healing is assessed using Simple Endoscopic Score for Cronh's Disease (SES-CD) score (0 or 1).
Rate of steroid-free remission | Up to 12 years
  Steroid-free remission is defined as weighted PCDAI < 12.5 or HBI <5 and no daily intake of prednisone (whatever the route). Rate of steroid-free remission will be described at each time point.
Proportion of participants with fistula remission (in participants with fistulizing CD at entry) | Up to 12 years
  Fistula remission is defined as closure for at least 2 consecutive visits of all fistulae that were draining at baseline
Change in Tanner's staging | From Month 0 to 12 years
  Tanner's staging is used to assess growth and pubertal development.
Proportion of participants with immunomodulator-free clinical remission at each time point | Up to 12 years
  The proportion of participants with immunomodulator-free clinical remission is assessed at each time point.
Incidence rate of infectious events | Up to 12 years
  The incidence rate of serious and non-serious opportunistic infections is assessed.
Incidence rate of all-cause hospitalizations | Up to 12 years
  Hospitalization will be determined from the health care utilization information.
Proportion of participants with steroid tapering at each time point (steroids daily dosing lower than at baseline) | Up to 12 years
  The proportion of participants with steroid tapering i.e., steroids daily dosing lower than at baseline (week 0) is assessed.
Change in height z-score | From Month 0 to 12 years
  Growth is assessed by monitoring changes in height z-score
Proportion of participants with CD-related surgery | Up to 12 years
  CD-related surgery includes subtotal colectomy with ileorectostomy, colectomy with ileo-anal pouch, Koch pouch, ileostomy, small bowel resection, and etc.
Incidence rate of CD- or drug-related hospitalizations | Up to 12 years
  Hospitalization will be determined from the health care utilization information.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (24):
- France (24):
  - Centre Hospitalier Lyon Sud /ID# 152667, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Hospitalier Lyon Sud /ID# 152668, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Hopital Clocheville /ID# 152831, Tours, Centre-Val de Loire
  - CHU de Besancon - Jean Minjoz /ID# 154197, Besançon, Doubs
  - Hopitaux de Brabois Adultes /ID# 152729, Vandœuvre-lès-Nancy, Lorraine
  - CHU Toulouse /ID# 153251, Toulouse, Occitanie
  - CHU Batiment Robert Debre /ID# 152665, Angers
  - CHU Bordeaux-Hopital Pellegrin /ID# 154620, Bordeaux
  - Chu de Bordeaux Hopital /Id# 157926, Bordeaux
  - Centre Hospitalier Universitai /ID# 155465, Caen
  - CHU Hopital d'Estaing /ID# 152664, Clermont-Ferrand
  - Hopital Jeanne de Flandre /Id# 155464, Lille
  - Hopital de la Timone /ID# 160133, Marseille
  - Hopital Jacques Monod /ID# 152663, Montivillier
  - Hopital de la Source /ID# 159947, Orléans
  - Hopital de la Source /ID# 165534, Orléans
  - Robert Debre Hopital, FR /ID# 152666, Paris
  - Hopital Armand Trousseau /Id# 152669, Paris
  - Hopital Armand Trousseau /Id# 157092, Paris
  - Necker Hopital, FR /ID# 152830, Paris
  - Chu Lyon Sud /Id# 152838, Pierre-Bénite
  - CHU de Rennes - Hospital Sud /ID# 152730, Rennes
  - Charles Nicolle Hosp chu rouen /ID# 152670, Rouen
  - Charles Nicolle Hosp chu rouen /ID# 158688, Rouen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/clinical-trials/adalimumab_P15-759.pdf